CLINICAL TRIAL: NCT00676819
Title: Comparison of the Pharmacodynamics and Pharmacokinetics of Insulin Aspart and Human Soluble Insulin in Geriatric Subjects With Type 2 Diabetes Mellitus
Brief Title: Comparison of the Pharmacodynamics and Pharmacokinetics of Insulin Aspart and Human Insulin in Elderly People With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ANA-1416
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin aspart
  Other Names: ANA; NovoRapid
Drug: human insulin

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate if the pharmacodynamic / pharmacokinetic properties of insulin aspart and human soluble insulin are different in elderly (65 years of age or older) with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Duration of diabetes for at least 12 months
* Current treatment with human insulin or insulin analogues for at least 6 months
* BMI equal to or below 35 kg/m2
* HbA1c equal to or greater than 10.0 %
* No clinically significant cardiovascular event as judged by the Investigator within the last 6 months prior to the study

Exclusion Criteria:

* History of any illness that, in the opinion of the Investigator might confound the results of the study or pose additional risk in administering the trial products to the subject
* Current treatment with systemic corticosteroids
* Any positive reaction of drug of abuse or alcohol screen
* Cardiac problems defined as: decompensated heart failure and/or angina pectoris
* Uncontrolled treated/untreated hypertension as judged by the Investigator or blood pressure > 180 mm Hg systolic and/or > 110 mm Hg diastolic
* Known or suspected allergy to trial product or related products
* Blood donation of more than 500 ml within the last 12 weeks
* The receipt of any investigational drug within 4 weeks prior to this trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2002-01-10 (Actual); Primary Completion 2002-07-19 (Actual); Study Completion 2002-07-19 (Actual)

PRIMARY OUTCOMES:
Glucose infusion rate | in the time period from 0 to 120 min after administration of trial products (AUCGIR(0-120 min))

SECONDARY OUTCOMES:
AUCGIR(0-300 min) the area under the GIR profile | in the interval 0-300 minutes post dosing
AUCGIR(0 min-end of clamp) the area under the GIR profile | in the interval 0-600 minutes post dosing (or 0 min until termination of the glucose clamp if abandoned early because of high blood glucose values)
AUCGIR(300min-end of clamp) the area under the GIR profile | in the interval 300-600 minutes post dosing (or 300 min until termination of the glucose clamp if abandoned early because of high blood glucose values)
GIRmax: the maximal GIR value | tmax, GIR: the time to maximal GIR value
early and late t50%, GIR | the time to early and late half-maximal GIR value
AUCINS(0-60 min) the area under the serum insulin (or serum insulin aspart) profile | in the interval 0-60 minutes post dosing
AUCINS(0-300 min) the area under the serum insulin (or serum insulin aspart) profile | in the interval 0-300 minutes post dosing
AUCINS(0min-end of clamp) the area under the serum insulin (or serum insulin aspart) profile | in the interval 0-600 minutes post dosing (or 0 min until termination of the glucose clamp if abandoned early because of high blood glucose values)
AUCINS(300min-end of clamp) the area under the serum insulin (or serum insulin aspart) profile | in the interval 300-600 minutes post dosing (or 300 min until termination of the glucose clamp if abandoned early because of high blood glucose values)
Cmax,ins: the maximal serum insulin (or serum insulin aspart) concentration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Cologne, Germany

REFERENCES:
- [Result] Krones R, Schutte C, Heise T. The rapid-acting properties of insulin aspart are preserved in elderly people with type 2 diabetes. Diabetes Obes Metab. 2009 Jan;11(1):41-4. doi: 10.1111/j.1463-1326.2008.00988.x. PMID 19120432
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com